CLINICAL TRIAL: NCT04107103
Title: A Study to Evaluate the Safety and Feasibility of the Combined Use of Nivolumab With Pemetrexed for the Treatment of Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Nivolumab Plus Pemetrexed for Head and Neck Squamous Cell Carcinoma
Acronym: NivoPlus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nivo Plus: IIT-0009
Record Dates: First submitted 2019-09-16; First posted 2019-09-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: SCCHN
MeSH Terms: interventions — Pemetrexed; Nivolumab

STUDY DESIGN:
Intervention Model Description: A single-arm, interventional study combining nivolumab with pemetrexed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): A single-arm combining nivolumab with pemetrexed
  Interventions: Drug: Combination Product: Nivolumab with Pemetrexed

INTERVENTIONS:
Drug: Combination Product: Nivolumab with Pemetrexed — Nivolumab 3 mg/kg IV q.2 weekly in combination with pemetrexed 500mg/m2 q.6weekly. Treatment with nivolumab will continue every 14-days, and pemetrexed treatment will continue every 42-days. Treatment continues until disease progression or toxicity resulting in treatment discontinuation or until 2 years of treatment.
  Other Names: Opdivo (trade name for Nivolumab); Alimta (brand name for Pemetrexed)

SUMMARY:
The purpose of this study is to find out what effects the combination of Nivolumab and Pemetrexed has on you and your cancer. The safety of this combination and the effectiveness of this treatment will be studied.

DETAILED DESCRIPTION:
The treatment of patients with SCCHN is challenging, and represents an area of high unmet need. Treatment options within this patient population are limited, and inadequately treated disease may cause high morbidity, negatively impacting quality of life and leading to increased costs for supportive care. To address the unmet needs of these patients, this exploratory trial combining pemetrexed with standard-of-care nivolumab, with an investigational plan to study clinical and health services outcomes is being proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients must have a diagnosis of histologically confirmed squamous cell carcinoma of the head and neck not amenable to curative intent therapy (surgery or radical chemoradiation).
3. Patients with squamous cell cancer of the head and neck (SCCHN) who either have a recurrence within 6 months of potentially curative neoadjuvant/adjuvant platinum-based therapy or recurrence after receiving plantium based therapy in a non-curative setting, and who have a good performance status. Nivolumab may also be considered for patients who are ineligible for a platinum-based chemotherapy.
4. Patients presenting with a diagnosis of HPV-related (p16+) squamous cell carcinoma without an unknown primary will be eligible for enrolment if the investigator deems a head and neck primary to be the most likely primary source.
5. Patients must be capable of providing consent to enrolment and treatment.
6. Patients with a performance status of ECOG 0-2(15) will be eligible for enrolment (see appendix 1).
7. Measurable disease must be present according to RECIST criteria V1.1(16) (see appendix 5).
8. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
9. Patients (men and women) of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 6 months after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

   * Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
10. Female patients who are breast-feeding should discontinue nursing prior to the first dose of study treatment and until 30 days after the last dose of study drug.
11. Male patients should agree to not donate sperm during the study and for a period of at least 6 months after last dose of study drug.
12. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
13. The following adequate organ function laboratory values must be met:

Hematological:

* Absolute neutrophil count (ANC) >1.5 x109/L
* Platelet count >100 x109/L
* Hemoglobin >9 g/dL (may have been transfused)

Renal:

-Estimated creatinine clearance ≥ 45 mL/min according to the Cockcroft-Gault formula (or l-ocal institutional standard method)

Hepatic:

* Total serum bilirubin <1.5x ULN
* AST and ALT <2.5x ULN (or ≤ 5 x ULN for patients with documented metastatic disease to the liver)

Exclusion Criteria:

1. History of pneumonitis requiring treatment with steroids.
2. History of active interstitial lung disease.
3. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
4. History of another malignancy or a concurrent malignancy;

   -Exceptions include patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ.
5. Active brain metastases or leptomeningeal disease.

   -Patients with treated brain metastases that are stable for 6 weeks will be eligible for enrolment.
6. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
7. Prior organ transplantation including allogeneic stem-cell transplantation.
8. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
9. Active infection requiring systemic therapy.
10. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAE v4.03 Grade ≥ 3).
11. Other severe acute or chronic medical conditions including inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
12. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 grade > 1); however, alopecia, sensory neuropathy ≤ grade 2, or other toxicities ≤ grade 2 not constituting a safety risk based on investigator's judgment are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 year after enrollment of last participant
  The number of participants who complete at least 2 cycles of combination nivolumab with pemetrexed for the treatment of advanced head and neck cancers, over the total duration of study.
Safety/tolerability (incidence of adverse events including immune related) | Through study completion up to 2 years
  Treatment related and non-related adverse events per CTCAE v.4.0.3 of nivolumab with pemetrexed for the treatment of advanced head and neck cancers. Incidence of adverse events, the number of dose modifications and discontinuations due to adverse events including immune-related adverse events.

SECONDARY OUTCOMES:
Response Rate | 1 year after enrollment of last participant.
  associated with combination nivolumab/pemetrexed therapy (defined as the proportion of participants achieving either a partial response or a complete response as best-overall response per RECIST criteria 1.1)
Progression free survival | 5 years from final study drug dose.
  associated with combination nivolumab/pemetrexed therapy (defined as the time between the date of treatment initiation and the date of disease progression or death (whatever the cause, whichever occurs first)
Overall Survival | 5 years from final study drug dose.
  associated with combination nivolumab/pemetrexed therapy. (Defined as the time between the date of treatment initiation and the date of death)
Patient reported quality of life | Through study completion, up to 2 years.
  associated with combination nivolumab/pemetrexed therapy (measured utilizing the Edmonton Symptom Assessment Score). This questionnaire includes six yes/no questions, 10 questions with a scale of 0 (no symptoms) to 10 (at the worst).

OTHER OUTCOMES:
Investigation of the role of CD71+ immature red blood cells in the response to treatment with immunotherapy | 1 year after last study drug dose.
  In this study the frequency of the CD71+erythrocyte cells' (blood draws at pre-chemo, post-chemo and post immunotherapy) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hatim Karachiwala, MD FRCPC, Principal Investigator — Alberta Health Services - Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Result] Emens LA, Middleton G. The interplay of immunotherapy and chemotherapy: harnessing potential synergies. Cancer Immunol Res. 2015 May;3(5):436-43. doi: 10.1158/2326-6066.CIR-15-0064. PMID 25941355
- [Result] Pivot X, Raymond E, Laguerre B, Degardin M, Cals L, Armand JP, Lefebvre JL, Gedouin D, Ripoche V, Kayitalire L, Niyikiza C, Johnson R, Latz J, Schneider M. Pemetrexed disodium in recurrent locally advanced or metastatic squamous cell carcinoma of the head and neck. Br J Cancer. 2001 Sep 1;85(5):649-55. doi: 10.1054/bjoc.2001.2010. PMID 11531245
- [Result] Gilbert J, Murphy B, Dietrich MS, Henry E, Jordan R, Counsell A, Wirth P, Yarbrough WG, Slebos RJ, Chung CH. Phase 2 trial of oxaliplatin and pemetrexed as an induction regimen in locally advanced head and neck cancer. Cancer. 2012 Feb 15;118(4):1007-13. doi: 10.1002/cncr.26364. Epub 2011 Jul 15. PMID 21766301
- [Result] Vermorken JB, Licitra L, Stohlmacher-Williams J, Dietz A, Lopez-Picazo JM, Hamid O, Hossain AM, Chang SC, Gauler TC. Phase II study of pemetrexed in combination with cisplatin and cetuximab in recurrent or metastatic squamous cell carcinoma of the head and neck. Eur J Cancer. 2013 Sep;49(13):2877-83. doi: 10.1016/j.ejca.2013.05.002. Epub 2013 May 30. PMID 23726971
- [Result] Davis M, Conlon K, Bohac GC, Barcenas J, Leslie W, Watkins L, Lamzabi I, Deng Y, Li Y, Plate JM. Effect of pemetrexed on innate immune killer cells and adaptive immune T cells in subjects with adenocarcinoma of the pancreas. J Immunother. 2012 Oct;35(8):629-40. doi: 10.1097/CJI.0b013e31826c8a4f. PMID 22996369
- [Result] Elahi S, Ertelt JM, Kinder JM, Jiang TT, Zhang X, Xin L, Chaturvedi V, Strong BS, Qualls JE, Steinbrecher KA, Kalfa TA, Shaaban AF, Way SS. Immunosuppressive CD71+ erythroid cells compromise neonatal host defence against infection. Nature. 2013 Dec 5;504(7478):158-62. doi: 10.1038/nature12675. Epub 2013 Nov 6. PMID 24196717
- [Result] Dunsmore G, Bozorgmehr N, Delyea C, Koleva P, Namdar A, Elahi S. Erythroid Suppressor Cells Compromise Neonatal Immune Response against Bordetella pertussis. J Immunol. 2017 Sep 15;199(6):2081-2095. doi: 10.4049/jimmunol.1700742. Epub 2017 Aug 4. PMID 28779022
- [Result] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Result] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- See also: ESC guidelines website — https://www.escardio.org/Guidelines/Clinical-Practice-Guidelines
- See also: AHA guidelines website — http://professional.heart.org/professional/GuidelinesStatements/UCM_492626_Guidelines-Statements-Search-Page.jsp